| Title | Implementation and evaluation of a post-diagnostic announcement protocol at the Neuroretinal Disease Reference Center RefeRet, Quinze-Vingts Hospital. |
|---|---|
| Acronyme | RP-DIAG |
| Principal Investigator | Pr Isabelle AUDO, CRMR |
| Sponsor | Quinze-Vingts National Vision Hospital (HNV des 15-20) |
| Study Justification | Retinitis pigmentosa (RP), the main genetic retinal dystrophy, affects approximately 1 in 4,000 people and is characterized by progressive vision loss. Receiving the diagnosis is often challenging: the long medical journey and lack of clear guidance increase anxiety sometimes leading to a break in follow-up care. Unlike in oncology, there are no established post-diagnosis recommendations in this field. The current process at the Quinze-Vingts National Vision Hospital is limited to a consultation with the ophthalmologist, without formal coordination of psychological or nurse support. The RP DIAG study aims to structure post-diagnosis follow-up (nurse and psychological support and to evaluate its feasibility, impact, and potential for long-term implementation and adaptation in other rare disease centers. |
| Study Objectives | <ol> <li>To evaluate a new post-diagnostic paramedical support pathway (nurse and psychological support) in order to improve care for patients with retinitis pigmentosa (RP).</li> <li>To collect data on patients' psychological experience after diagnosis using the Hospital Anxiety and Depression Scale (HADS).</li> <li>To assess the feasibility of generalizing the support pathway, including the workload for clinical teams, using the RETEX questionnaire, and to provide the basis for a standardized, sustainable post-diagnostic protocol that could potentially be reproduced in other ophthalmology rare disease centers.</li> </ol> |
| Study Category and Type | Pilot study, RIPH2 category. Randomized, prospective, longitudinal, monocentric comparative study. |
| Evaluation Criteria and Outcome Measures | <ol> <li>Patient-perceived satisfaction: Measured using the PREM (Patient-Reported Experience Measure) questionnaire, comparing: <ul> <li>An experimental group receiving the structured nurse/psychological follow-up</li> <li>A control group receiving usual care</li></ul></li></ol> |
| Inclusion Criteria | <ul> <li>quantitatively evaluate the benefits of the intervention.</li> <li>Diagnosed with retinitis pigmentosa and receiving care at the Rare Disease Reference Center (CRMR), with diagnosis disclosure occurring after the project's initiation.</li> <li>Aged between 18 and 65 years.</li> <li>Male or female.</li> <li>French-speaking.</li> <li>Has a valid telephone number.</li> <li>Resident of France</li> </ul> |
| Exclusion Criteria | <ul> <li>Resident of France.</li> <li>Individuals enrolled in a therapeutic clinical trial (for 12 months)</li> <li>Individuals deprived of liberty by judicial or administrative decision (art. L1121-6 of the French Public Health Code)</li> <li>Adults under legal protection measures or unable to provide consent (art. L1121-8 of the French Public Health Code)</li> <li>Individuals with other medical conditions or taking treatments likely to interfere with study assessments</li> <li>Participants unable to attend all study visits</li> </ul> |

| | T | | | | |
|---|---|---|---|---|---|
| | - Pregnant, postpartum, or breastfeeding women (according to art. L1121-5 of the French Public Health Code). | | | | |
| Criteria for early<br>withdrawal or study<br>discontinuation | <ul> <li>Occurrence of other medical conditions or treatments which could interfere with the planned assessments of the study;</li> <li>A participant may decide at any time to withdraw from the study;</li> <li>A participant may also be withdrawn from the study by the investigator.</li> </ul> | | | | |
| Constraints and Risks | This pilot study does not present any foreseeable medical risks. | | | | |
| Population | Target population: Adult patients diagnosed with retinitis pigmentosa (RP) who meet the inclusion criteria – first encounter with the name of their condition. Sample: 80 patients (40 in the experimental group, 40 in the control group). Randomization: Performed using the RedCAP software. | | | | |
| Study Procedure | Experimental Group | Experimental Group (n=40) | | | |
| | <ol> <li>Visit 1 (Diagnosis Announcement): Ophthalmologist consultation; project information; optional initial discussion with the nurse.</li> <li>Consent Collection</li> <li>Visit 2 (Day 15): Nurse consultation (in-person or by phone, ~1 hour) to explain the disease and procedures, and assess emotional state (HADS-1).</li> <li>Visit 3 (6 months): Nurse consultation (HADS-2); psychologist consultation offered.</li> <li>Visit 4 (12 months): Ophthalmology consultation; nurse consultation (HADS-3); PREM questionnaire to assess patient satisfaction.</li> <li>Control Group (n=40) <ul> <li>Usual care: Diagnosis consultation followed by a 12-month follow-up visit. At the 12-month visit, the patient completes the PREM questionnaire. No systematic nurse or psychological follow-up between diagnosis and the 12-month visit, unless requested by the patient.</li> </ul> </li> <li>Visit Schedule Summary</li> </ol> | | | | |
| | Visits | Day 0 | Day 15 | 6 Months | 12 Months |
| | Visits | (Announcement) | (V1) | (V2) | (V3) |
| | Informed Consent | X | | - | - |
| | Control Group<br>(Usual Care) | PREM | - | - | PREM |
| | Experimental<br>Group (Enhanced<br>Support) | HADS | HADS | HADS +<br>Psychologist | HADS +<br>PREM |
| Planned Study Timeline | Expected study start date: September 2025 Participant involvement duration: 12 months Visit frequency: As detailed in the visit schedule above Expected inclusion period: 10 months (approximately 8 patients enrolled per month) Total study duration: 24 months | | | | |
| | Total study duration | : 24 months | | | |
| Source of Funding | Total study duration The project is funded | | ram of the GI | IRCL | |